CLINICAL TRIAL: NCT05770193
Title: Effect Of Kinesio Tape Versus Diaphragmatic Breathing Exercise In Post COVID-19 Patients(A Comparative Study)
Brief Title: Effect of Kinesio Tape Versus Diaphragmatic Breathing Exercise In Post COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdallah Salah Abdallah Gabr, B.Sc. in Physical Therapy Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004370
Record Dates: First submitted 2023-03-10; First posted 2023-03-15 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Post COVID-19 Condition
Keywords: Kinesio tape; Diaphragmatic breathing exercise; Post COVID-19; six-minute walk test; Oxygen Saturation; Fatigue Severity Scale; Quality of life
MeSH Terms: interventions — Cognitive Behavioral Therapy; Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pursed lip breathing and CBT in addition to kinesio tape. (Experimental): patients will receive pursed lip breathing and cognitive-behavioral therapy in addition to kinesio tape.
  Interventions: Other: Pursed lip breathing; Other: Cognitive Behavior Therapy; Other: Kinesio tape
- pursed lip breathing and CBT in addition to diaphragmatic breathing exercise. (Experimental): patients will receive pursed lip breathing and cognitive-behavioral therapy in addition to diaphragmatic breathing exercise
  Interventions: Other: Pursed lip breathing; Other: Cognitive Behavior Therapy; Other: Diaphragmatic breathing exercise
- pursed lip breathing and CBT. (Active Comparator): patients will receive pursed lip breathing and cognitive-behavioral therapy.
  Interventions: Other: Pursed lip breathing; Other: Cognitive Behavior Therapy

INTERVENTIONS:
Other: Pursed lip breathing — The position for every patient will be long sitting, and then he will be instructed to breathe in through the nose for 2 seconds. Purse the lips as if about to blow out the candles on a cake. Breathe out very slowly through pursed lips for 4 to 6 seconds, and then repeat for 5 to 10 minutes. The intervention will be done two days a week, through six weeks for all participants by a physiotherapist.
Other: Cognitive Behavior Therapy — A structured, 6-session psycho-therapeutic intervention, occurring once weekly, will be performed According to the CBT session structure provided by Cully and Teten, with some modifications, Each session will be approximately 1 hour.
  Other Names: (CBT)
Other: Diaphragmatic breathing exercise — The patient will lie in supine position, and then he will be asked to rest for 5 min and lay on their back on a flat surface with pillows under their head and knees for support. One hand will be placed on the abdomen and the other on the upper part of the chest wall. When inhaling, the hand on the abdomen will move upward, while the other hand will remain as still as possible. When exhaling, the hand on the abdomen will move downwards, while the other hand will remain as still as possible again. Breathing will be performed quickly, deeply and without causing tiredness. The breaths should be inhaled through the nose and exhaled through the mouth.
  The diaphragmatic breathing exercise will consist of three sets of 10 repetitions, with 30 seconds of rest between each set
  Arms: pursed lip breathing and CBT in addition to diaphragmatic breathing exercise.
Other: Kinesio tape — The position for every patient will be sitting during application of the tape. The diaphragm muscle will be covered with kinesio tape both anteriorly and posteriorly along the subcostal region. Anteriorly, the base point of an "I" shaped kinesio tape will be applied on xiphoid process with 50_75% tension on the linea Alba and the tails of the tape were applied toward subcostal curvature. Posteriorly, a second "I" shaped Kinesio Tape will be applied from the back The base point of the tape will be applied on the projection of 12th Thoracic vertebra with 50 _75% tension and the tails will be applied toward the ribs.
  Arms: pursed lip breathing and CBT in addition to kinesio tape.

SUMMARY:
According to WHO, current evidence suggests some people experience a variety of long-term effects after they recover from their initial illness. These effects are collectively known as post COVID-19 condition or "long COVID. While most people who develop COVID-19 fully recover, some people develop effects like fatigue, breathlessness, functional activities and cognitive dysfunction. At present, there is no specific medication therapy for people with post COVID-19 condition.

DETAILED DESCRIPTION:
Lungs are the main organs affected by the virus so many respiratory complications occur, like increasing breathing effort marked by the usage of auxiliary respiratory muscle and paradoxical breathing pattern. However, when a patient with the corona virus become negative, the symptoms during Covid-19 infection do not immediately disappear, these symptoms can even continue for months. A study on Long Covid stated that, about 87.4% of people reported feeling at least one persistent symptom and the most common was chronic fatigue and shortness of breath. Physiotherapy rehabilitation, such as breathing exercises and chest physiotherapy, can be effective adjuvant therapies in COVID-19 patients. Different therapies are suggested to treat Covid-19 complications as Pursed lip breathing exercise which is effective in improving respiratory rate and reducing dyspnea in Covid-19 patients.

Cognitive Behavior Therapy (CBT) has a great impact in promoting the physical and psychological health of patients during COVID-19.

A series of recent studies has indicated that, a telerehabilitation program consisting of 1-week respiratory exercises was found to be effective, safe, and feasible in Covid-19 patients with mild to moderate symptomatology. A recent study by Cascella et al. concluded that, breathing exercises and chest therapy can be used to help post COVID-19 patients regain their normal breathing capacity.

kinesio tape helps with neuromusculoskeletal rehabilitation by activating cutaneous mechanoreceptors, which interact with deeper tissues via continuous sensory and mechanical stimuli in the skin, forming a neural arc and proper motor response. In patients with COPD, Kinesio tape combined with deep breathing exercises significantly improved pulmonary function, perceived severity of dyspnea, and fatigue, and had a positive effect on functional capacity.

Desai et al. concluded in their study that, kinesio tape applied to the diaphragm has a good prognosis for diaphragm muscle weakness. It improved maximum inspiratory pressure and diaphragmatic excursion range.

60 Patients will be assignment randomly into three groups: Group A: 20 patients will receive pursed lip breathing and cognitive-behavioral therapy in addition to kinesio tape.

Group B: 20 patients will receive pursed lip breathing and cognitive-behavioral therapy in addition to diaphragmatic breathing exercise.

Group C: 20 patients will receive pursed lip breathing and cognitive-behavioral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. People who have a history of probable or confirmed SARS-CoV-2 infection; usually within three months from the onset of COVID-19, with symptoms and effects that last for at least two months.
2. Aged 18-45 years old.
3. Non-hospitalized.
4. Both sexes will be included.
5. Body mass index (BMI) range from (18.5 to 24.9 kg/m2).
6. Patients with low to moderate physical activity, according to the International Physical Activity Questionnaire (IPAQ) Arabic version.
7. Patients with grade 2 or higher on Modified Medical research council (Dyspnea Scale).
8. Able to read and write.
9. Willing and able to complete study procedures. -

Exclusion Criteria:

* 1. Patients on medications that would influence exercise performance such as beta-blockers or antiretroviral therapy.

  2. Enrolled in another interventional clinical research trial in the previous 30 days.

  3. Pregnancy. 4. Had significant hepatic or renal dysfunction. 5. New onset of arrhythmia and myocardial ischemia. 6. Hospitalized. 7. Cardiac disease, chronic respiratory disease, active infection, severe endocrine or metabolic diseases.

  8. Cognitive impairment. 9. Patients with red flag indicators such as chest pain, critical drop in oxygen saturation, musculoskeletal or neurologic limitations, and unconscious patients.

  10. Contraindications of using kinesio tape as Malignancy, Infection, cellulitis, Open Wound, DVT, and Previous allergic reaction to kinesio tape

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-11 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Modified Medical research council | 6 weeks
  It will used to assess Dyspnea, This test is very easy to perform; it is valid and correlates with clinical parameters and parameters of respiratory function.

SECONDARY OUTCOMES:
Pulse oximeter | 6 weeks
  It will be used to measure oxygen saturation. It is a valid tool to measure oxygen saturation. Powers et al, concluded that Pulse oximeter is useful tool in estimating percent arterial oxygen saturation of hemoglobin in healthy subjects.
  It will be attached to the thump and the reading will be recorded
Arabic version of The Fatigue Severity Scale | 6 weeks
  It will be used to measure fatigue level. The FSS showed satisfactory reliability and validity and thus can be regarded as a feasible measure of self-reported fatigue.
  In addition to measuring the presence and degree of fatigue in a sample of Arabic patients, the Arabic version of the FSS also shown indications of internal consistency, relative test-retest reliability, and construct validity, supporting its application in clinical practice and research.
six-minute walk test | 6 weeks
  It will be used to measure physical or functional performance. The 6-min walk is a reliable and valid measure of physical endurance in older adults and it moderately reflects overall physical functional performance.
  A newer application of the six-minute walk test is noted for patients who have had COVID-19 pneumonia with prolonged respiratory symptoms.
The World Health Organization Quality-of-Life Scale (WHOQOL-BREF). | 6 weeks
  The World Health Organization Quality-of-Life Scale (WHOQOL-BREF) provides a reliable, valid, and brief assessment of quality-of-life.
  The Arabic translation of the WHOQOL-BREF has impressive reliability and validity indices. There will be a four-domain score. The four domain scores will denote an individual perception of quality of life in each particular domain. Domain scores are scaled in a positive direction higher scores denote higher quality of life. The mean score of items within each domain is used to calculate the domain score. Mean scores are then multiplied by 4 in order to make domain scores comparable with the scores used in the WHOQOL-100

CONTACTS AND LOCATIONS:
Overall Officials: fatma S Amin, Principal Investigator — Professor of Basic Science / Faculty of Physical therapy/ Cairo university; Doaa A Elimy, Principal Investigator — Lecturer of Basic Science /Faculty of Physical therapy/ Cairo university; Ahmed A mohamed, Principal Investigator — Professor of chest disease Faculty of medicine banha university
Locations (1):
- Abdallah salah abdallah gbr, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Study protocol